CLINICAL TRIAL: NCT00010166
Title: Phase II Trial Of Adjuvant 2'2'-Difluoro-2'-Deoxycytidine (Gemcitabine) And External Beam Radiation For The Treatment Of Resectable Pancreatic Cancer
Brief Title: Gemcitabine and Radiation Therapy in Treating Patients With Cancer of the Pancreas
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: REBACDR0000068452; CCCWFU-57198; NCI-104
Record Dates: First submitted 2001-02-02; First posted 2003-01-27 (Estimated); Last update posted 2021-09-09 (Actual); Status verified 2021-09

CONDITIONS: Pancreatic Cancer
Keywords: stage I pancreatic cancer; adenocarcinoma of the pancreas
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine; Chemotherapy, Adjuvant; Radiotherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Drug: gemcitabine hydrochloride
Procedure: adjuvant therapy
Radiation: radiation therapy

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to damage tumor cells. Gemcitabine may make tumor cells more sensitive to radiation therapy. Combining chemotherapy with radiation therapy after surgery may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combining gemcitabine with radiation therapy in treating patients who have undergone surgery to remove cancer of the pancreas.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the time to disease progression, local control, and survival of patients with previously resected pancreatic cancer treated with adjuvant gemcitabine and radiotherapy.

OUTLINE: This is a multicenter study.

Patients receive gemcitabine IV over 30-60 minutes on days 1, 4, 8, 11, 15, 18, 22, 25, 29, and 32 and undergo radiotherapy on days 1-5, 8-12, 15-19, 22-26, 29-33, and 36-38 in the absence of disease progression or unacceptable toxicity.

Beginning at least 4 weeks after chemoradiotherapy, patients without disease progression and with less than 10% weight loss during study receive additional gemcitabine IV over 30 minutes on days 1, 8, and 15. Treatment repeats every 28 days for a total of 2 courses.

Patients are followed every 8 weeks for 6 months and then every 3 months for up to 2 years.

PROJECTED ACCRUAL: A total of 72 patients will be accrued for this study within 2.2 or 3.4 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed invasive adenocarcinoma of the pancreas

  * Prior gross total resection via a pancreaticoduodenectomy (Whipple resection or total pancreatectomy) within the past 2 months
* No clinical evidence of gross residual disease at time of surgery

  * No focally positive margins (tumor at the margin)
* No unresected nodal disease or metastatic disease to the liver, peritoneal surfaces, or elsewhere

PATIENT CHARACTERISTICS:

Age:

* Over 18

Performance status:

* ECOG 0-2

Life expectancy:

* More than 6 months

Hematopoietic:

* Granulocyte count greater than 1,500/mm3
* Hemoglobin greater than 10 g/dL
* Platelet count greater than 100,000/mm3

Hepatic:

* Bilirubin less than 2.0 mg/dL

Renal:

* Creatinine less than 2.0 mg/dL

Other:

* Able to maintain adequate oral nutrition
* Documented stable weight (no more than 5 lbs weight loss) for at least 2 weeks prior to study
* No other malignancy within the past 2 years except inactive nonmelanoma skin cancer or carcinoma in situ of the cervix or breast
* Non-metastatic prostate cancer allowed if more than 2 year survival likely
* No other serious medical or psychiatric illness that would preclude study or limit survival to less than 2 years
* Not pregnant
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No concurrent routine growth factors

Chemotherapy:

* No prior chemotherapy for pancreatic cancer

Endocrine therapy:

* Not specified

Radiotherapy:

* No prior abdominal radiotherapy for pancreatic cancer

Surgery:

* See Disease Characteristics

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2000-12-01 (Actual); Primary Completion 2003-10-03 (Actual); Study Completion 2003-10-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arthur William Blackstock, MD, Study Chair — Wake Forest University Health Sciences
Locations (1):
- Comprehensive Cancer Center at Wake Forest University, Winston-Salem, North Carolina, United States

REFERENCES:
- [Result] Blackstock AW, Mornex F, Partensky C, Descos L, Case LD, Melin SA, Levine EA, Mishra G, Limentani SA, Kachnic LA, Tepper JE. Adjuvant gemcitabine and concurrent radiation for patients with resected pancreatic cancer: a phase II study. Br J Cancer. 2006 Aug 7;95(3):260-5. doi: 10.1038/sj.bjc.6603270. Epub 2006 Jul 25. PMID 16868545